CLINICAL TRIAL: NCT03512561
Title: Impact of the Presurgical Visit of Nursing on the Well-being of the Patient Before a Surgical Process at the Parc Taulí Health Corporation.
Brief Title: Impact of the Presurgical Visit of Nursing on the Well-being of the Surgical Patient.
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Francisco Zamora Carmona, Nursing, Corporacion Parc Tauli
Other Study IDs: EST-VPI-2017
Record Dates: First submitted 2018-03-08; First posted 2018-04-30 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Nurse's Role; Preoperative Care; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
.A surgical intervention involves the participant and his / her family in a very stressful situation with a biopsychosocial alteration of the participant, often presenting a lack of knowledge of the surgical process from admission to hospital discharge. Researchers (nursing) began to make prior visits to the surgical procedure to reduce anxiety and provide information about the surgical process. The importance of the presurgical nursing visit (PNV) is sought, how to achieve a better health education throughout the surgical process, improve communication between professionals through standardized records, contributing to an optimal approach to the participant, increasing well-being, health and the satisfaction of the participant

DETAILED DESCRIPTION:
In our Center, PNVs are carried out in the Ambulatory Area (External Consultations) in a specific and personalized nursing consultation, within an established and multidisciplinary program. One week before surgery, the patient and a family / primary caregiver are cited.

The PNV conducts a semi-structured interview; the content may vary according to the type of surgery, but in general it can be understood as all those nursing interventions; how to provide information, support, advice and training to the patient and his family (primary caregiver).

It is an innovative experience since it has been carried out for a short time. The PNV have been gradually restructured and continue to grow, since their establishment has been positively valued in the different services thanks to the experience gained and the numerous bibliographic references that demonstrate the beneficial results for the patient and the health system.

A total of 356 participants have been calculated (surveys answered in more than 3 months), taking into account an approximate population of 1,172 programmed interventions carried out in 1 year, with a confidence interval of 95%, accuracy of 3% a proportion of 5% and with an expected loss of 15%.

Sample:

Arthralplasia of knee / hip N 480 n 92 Cystectomies N 24 n 19 Esophagogastric with coloplasty N 24 n 19 Hysterectomy N 24 n 19 Colon / rectum N 192 n 65 Lumpectomy with sentinel lymph nodes N 222 n 74 Caesarean section N 206 n 68

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone the pre-surgical nursing visit (personalized).
* Patients over 18 years of age
* Live accompanied and / or with own resources of help.
* Having signed the informed consent.

Exclusion Criteria:

* Not having signed the informed consent.
* Not having done the questionnaires after pre-surgical nursing visit (STAI, EQ-5D-5L)
* For surgical complications that do not allow the telephone survey, or focal groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients who are going to be operated
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
The participant is satisfied throughout the surgical process, in relation to information, health education and personalized attention to the presurgical nursing visit (PNV) | 3 months
  Number of participants who are satisfied with the experience of the surgical procedure and if this is what is explained in the presurgical nursing visit, for the evaluation of the importance of the visit in the surgical process.

SECONDARY OUTCOMES:
The participant feels well-being due to the care received by the professionals throughout the surgical process. | 3 month
  Number of participants who perceive welfare linked to the quality of care of the surgical process.
The participant has preoperative and postoperative anxiety in more than three months, relating it to the information provided in the presurgical nursing visit. | 3 months
  Number of participants who perceive pre and postsurgical anxiety and if it is linked to the information provided during the visit.
The participant perceives better quality of presurgical and postoperative life in more than three months; in relation to the training given during the pre-surgical nursing visit. | 3 months
  Number of participants who perceive an improvement in the quality of life and if it is linked to the information provided during the visit.

CONTACTS AND LOCATIONS:
Overall Officials: Francesc Zamora-Carmona, Nurse, Principal Investigator — Corporacion Parc Tauli
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No